CLINICAL TRIAL: NCT04855162
Title: Use of Lung Ultrasound in Evaluating Physiological Response to Awake Self Proning
Status: Completed | Type: Observational
Sponsor: Rush University Medical Center (Other)
Collaborators: Hospital Civil de Guadalajara (Other)
Responsible Party: Principal Investigator, Jie Li, Associate Professor, Rush University Medical Center
Other Study IDs: 21040601
Record Dates: First submitted 2021-04-13; First posted 2021-04-22 (Actual); Last update posted 2021-11-15 (Actual); Status verified 2021-11

CONDITIONS: Covid19
Keywords: Awake prone; Self prone
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary objective of this study is to explore the physiological mechanism of awake, self proning among patients with acute hypoxemic respiratory failure induced by COVID-19, using LUS in the first three days and explore the predictive value of LUS in patients' outcome.

DETAILED DESCRIPTION:
Lung ultrasound (LUS) has recently gained popularity among the imaging methods to perform bedside assessment of critically ill patients to guide clinical management. LUS is a non-invasive and easy-to-perform procedure that provides precise data on lung aeration, lung recruitment, lung morphology, and lung perfusion. Studies have shown that LUS is a useful tool in monitoring lung reaeration in intubated patients diagnosed with traditional ARDS undergoing prone positioning; however there are mixed findings in terms of the use of LUS in predicting potential prone positioning response. A recent study found that the non-intubated COVID-19 patients who responded to prone positioning had more pronounced disturbances of aeration in posterior regions, however, they only investigated patients' response to the first prone positioning and the information for the patients' outcome is lacking. In our previous study with intubated COVID-19 patients, we found that patients' response to the subsequent prone positioning had higher predictive value than the response to the first prone positioning. Therefore, the primary objective of this study is to explore the physiological mechanism of awake, self proning among patients with acute hypoxemic respiratory failure induced by COVID-19, using LUS in the first three days and explore the predictive value of LUS in patients' outcome.

ELIGIBILITY:
Inclusion Criteria:

1. Adult subjects 18 years and older,
2. Confirmed COVID-19 diagnosis
3. Acute hypoxemic respiratory failure (SpO2/FiO2 or PaO2/FiO2 <300)
4. Ordered self-prone positioning per medical team

Exclusion Criteria:

1. Pregnant
2. Palliative care

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients with acute hypoxemic respiratory failure due to COVID-19 who are admitted at Rush University Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2021-07-21 (Actual); Primary Completion 2021-10-07 (Actual); Study Completion 2021-10-23 (Actual)

PRIMARY OUTCOMES:
SpO2/FiO2 pre prone in day 1 | pre prone in day 1
  Patients' response of oxygenation using SpO2/FiO2
SpO2/FiO2 post prone in day 1 | post prone in day 1
  Patients' response of oxygenation using SpO2/FiO2
SpO2/FiO2 pre prone in day 2 | Pre prone in day 2
  Patients' response of oxygenation using SpO2/FiO2
SpO2/FiO2 post prone in day 2 | Post prone in day 2
  Patients' response of oxygenation using SpO2/FiO2
SpO2/FiO2 pre prone in day 3 | Pre prone in day 3
  Patients' response of oxygenation using SpO2/FiO2
SpO2/FiO2 post prone in day 3 | Post prone in day 3
  Patients' response of oxygenation using SpO2/FiO2
Lung Ultrasound Score pre prone in day 1 | Pre prone in day 1
  Patients' response of oxygenation using Lung ultrasound score
Lung Ultrasound Score post prone in day 1 | Post prone in day 1
  Patients' response of oxygenation using Lung ultrasound score
Lung Ultrasound Score pre prone in day 2 | Pre prone in day 2
  Patients' response of oxygenation using Lung ultrasound score
Lung Ultrasound Score post prone in day 2 | Post prone in day 2
  Patients' response of oxygenation using Lung ultrasound score
Lung Ultrasound Score pre prone in day 3 | Pre prone in day 3
  Patients' response of oxygenation using Lung ultrasound score
Lung Ultrasound Score post prone in day 3 | Post prone in day 3
  Patients' response of oxygenation using Lung ultrasound score

CONTACTS AND LOCATIONS:
Overall Officials: Jie Li, Principal Investigator — Rush University
Locations (2):
- Rush University Medical Center, Chicago, Illinois, United States
- Hospital Civil Fray Antonio Alcalde, Guadalajara, Jalisco, Mexico

REFERENCES:
- [Background] Langer T, Brioni M, Guzzardella A, Carlesso E, Cabrini L, Castelli G, Dalla Corte F, De Robertis E, Favarato M, Forastieri A, Forlini C, Girardis M, Grieco DL, Mirabella L, Noseda V, Previtali P, Protti A, Rona R, Tardini F, Tonetti T, Zannoni F, Antonelli M, Foti G, Ranieri M, Pesenti A, Fumagalli R, Grasselli G; PRONA-COVID Group. Prone position in intubated, mechanically ventilated patients with COVID-19: a multi-centric study of more than 1000 patients. Crit Care. 2021 Apr 6;25(1):128. doi: 10.1186/s13054-021-03552-2. PMID 33823862
- [Background] Wang XT, Ding X, Zhang HM, Chen H, Su LX, Liu DW; Chinese Critical Ultrasound Study Group (CCUSG). Lung ultrasound can be used to predict the potential of prone positioning and assess prognosis in patients with acute respiratory distress syndrome. Crit Care. 2016 Nov 30;20(1):385. doi: 10.1186/s13054-016-1558-0. PMID 27899151
- [Background] Avdeev SN, Nekludova GV, Trushenko NV, Tsareva NA, Yaroshetskiy AI, Kosanovic D. Lung ultrasound can predict response to the prone position in awake non-intubated patients with COVID-19 associated acute respiratory distress syndrome. Crit Care. 2021 Jan 25;25(1):35. doi: 10.1186/s13054-021-03472-1. No abstract available. PMID 33494771
- [Result] Weiss TT, Cerda F, Scott JB, Kaur R, Sungurlu S, Mirza SH, Alolaiwat AA, Kaur R, Augustynovich AE, Li J. Prone positioning for patients intubated for severe acute respiratory distress syndrome (ARDS) secondary to COVID-19: a retrospective observational cohort study. Br J Anaesth. 2021 Jan;126(1):48-55. doi: 10.1016/j.bja.2020.09.042. Epub 2020 Oct 10. PMID 33158500
- [Derived] Ibarra-Estrada M, Gamero-Rodriguez MJ, Garcia-de-Acilu M, Roca O, Sandoval-Plascencia L, Aguirre-Avalos G, Garcia-Salcido R, Aguirre-Diaz SA, Vines DL, Mirza S, Kaur R, Weiss T, Guerin C, Li J. Lung ultrasound response to awake prone positioning predicts the need for intubation in patients with COVID-19 induced acute hypoxemic respiratory failure: an observational study. Crit Care. 2022 Jun 27;26(1):189. doi: 10.1186/s13054-022-04064-3. PMID 35761404